CLINICAL TRIAL: NCT05641220
Title: Biopsy Versus Resection in Elderly Glioblastoma Patients. A Prospective Cohort Study.
Acronym: BIOPSY
Status: Not yet recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, A.J.P.E. VIncent, Prof. Dr., Erasmus Medical Center
Other Study IDs: MEC-2022-0678
Record Dates: First submitted 2022-11-18; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; High grade glioma; Surgical management; Biopsy; Resection
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Biopsy: Newly diagnosed elderly (>70 years of age) glioblastoma patients who undergo biopsy
- Resection: Newly diagnosed elderly (>70 years of age) glioblastoma patients who undergo resection

SUMMARY:
This trial is set up as a prospective observational cohort study to identify if either biopsy or resection should be the surgical modality of choice in elderly glioblastoma patients with a newly diagnosed tumor. Patients who are considered eligible for GBM resection or biopsy will be included. Through shared-decision making patients and their treating physicians will decide upon resection or biopsy. Written informed consent will be obtained. Participants will be followed for 1 year postoperative to assess potential differences in health-related quality of life and overall survival.

Follow-up will consist of health-related quality of life questionaires and neurological assessment at 6 weeks, 3 months, 6 months and 12 months postoperative. Additionally Cognitive and neuro-linguistic tests will be done at 3 months postoperative. These will be compared to results pre-operative.

After surgery, patients will receive standard adjuvant treatment with concomitant Temozolomide and radiation therapy, and standard follow-up. Patients in whom the diagnosis GBM is not confirmed in histological analyses will be excluded from the study. Total study duration will be 4 years, of which 3 years will comprise patient inclusion, with a follow-up duration of 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥70 years
2. Tumor diagnosed as glioblastoma on MRI with distinct ring-like pattern of contrast enhancement with thick irregular walls and a core area reduced signal suggestive of tumor necrosis as assessed by the surgeon.
3. Karnofsky Performance Score (KPS) ≥70
4. Written Informed consent

Exclusion Criteria:

1. Tumors of the cerebellum, brain stem or midline
2. Multifocal contrast enhancing lesions
3. Substantial non-contrast enhancing tumor areas suggesting low grade gliomas with malignant transformation
4. Medical reasons precluding MRI (e.g. pacemaker)
5. Inability to give consent as assessed by neurosurgeon (e.g. language barrier)
6. Severe aphasia prohibiting neurolinguistic testing and comprehension of informed consent
7. Previous brain tumor surgery
8. Previous low-grade glioma
9. Second primary malignancy within the past 5 years with the exception of adequately treated in situ carcinoma of any organ or basal cell carcinoma of the skin.

Ages: 70 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adults with presumed Glioblastoma on first diagnostic MRI-scan.
Sampling Method: Probability Sample
Enrollment: 325 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 12 months
  Defined as the time from diagnosis to the death of the patient from any cause
The difference in mean change score of physical functioning, as measured with the EORTC QLQ-C30 physical functioning scale, between the two groups at 6 weeks and 3 months after surgery compared to mean score on baseline | 6 weeks and 3 months after surgery
  Measured with the European Organisation for Research and Treatment of Cancer Core Quality of Life questionnaire (EORTC QLQ-C30), a higher scores means a worse outcome. We assume a minimally important difference of 7 between the 2 groups.

SECONDARY OUTCOMES:
Progression-free survival (PFS), defined as the time from diagnosis to disease progression | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months after surgery
  Increase in residual tumor volume of more than 25%, or occurrence of a new tumor lesion with a volume greater than 0.175cm3), or death. As according to the RANO criteria.
The difference in mean change score of physical functioning, as measured with the EORTC QLQ-C30 physical functioning scale, between the two groups at 6 months and 12 months after surgery compared to mean score on baseline. | at 6 months and 12 months after surgery
  Measured with the European Organisation for Research and Treatment of Cancer Core Quality of Life questionnaire (EORTC QLQ-C30), a higher scores means a worse outcome.
The proportion of patients with deterioration, improvement or stable physical functioning, as measured with the EORTC QLQ-C30 physical functioning scale at 6 weeks and 3 months compared to baseline. | 6 weeks and 3 months after surgery
  Measured with the European Organisation for Research and Treatment of Cancer Core Quality of Life questionnaire (EORTC QLQ-C30), a higher scores means a worse outcome.
Descriptive reporting of changes in the mean scores on the other health-related quality of life (HRQoL) scales at 6 weeks and 3 months after surgery. | at 6 weeks and 3 months postoperative
  HRQoL will be measured using the Measured with the European Organisation for Research and Treatment of Cancer (EORTC) Core Quality of Life questionnaire (QLQ-C30), EORTC , EORTC brain cancer module (QLQ-BN20) and EuroQol 5 Dimensions (EQ-5D) questionnaires. A higher scores means a worse outcome.
Proportion of patients with NIHSS (National Institute of Health Stroke Scale) deterioration, improvement or stability at 6 weeks and 3 months after surgery | at 6 weeks and 3 months postoperative
  In which deterioration is defined as an increase of at least one point and improvement as a decrease of at least one point on the total NIHSS score compared to this score at baseline.
Descriptive reporting of differences between the groups in cognitive and neuro-linguistic screening at 3 months compared to baseline. | 3 months postoperative
  as measured by the Aphasia Bedside Check (ABC), Shortened Token Test, verbal fluency (category and letter), Montreal Cognitive Assessment (MOCA) and optionally CAT-NL Picture Description and Object Naming.
Comparison of the (S)AEs in both groups. | 6 weeks postoperative
Cost-effectiveness between the two treatments. | 12 months postoperative
  Measured as total intramural medical costs, for a 1 year time horizon

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud J.P.E. Vincent, Prof. Dr., Principal Investigator — Erasmus MC, department of neurosurgery
Locations (6):
- Netherlands (6):
  - Northwest Clinics, Alkmaar
  - Medical Spectrum Twente, Enschede
  - Maastricht UMC, Maastricht
  - Erasmus MC, Rotterdam
  - Haaglanden MC, The Hague
  - Elisabeth-TweeSteden Hospital, Tilburg

IPD SHARING:
Plan to Share IPD: Undecided